CLINICAL TRIAL: NCT06193031
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Single Ascending Dose Study of C16TR for Inhalation to Determine Its Safety, Tolerability, and Pharmacokinetics With an Open-label Tyvaso® Cohort in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of C16TR for Inhalation With Tyvaso® Cohort in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INS1009-101
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — hexadecyl-treprostinil; treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Tyvaso®+C16TR Dose A or Tyvaso®+Placebo (Experimental): Participants received a single dose of Tyvaso® on Day 1, then randomized to receive either a single dose of C16TR for inhalation (Dose A) or matching placebo on Day 2 in Cohort 1.
  Interventions: Drug: C16TR; Drug: Placebo; Drug: Tyvaso®
- Cohort 2: C16TR Dose B or Placebo (Experimental): Participants were randomized to receive a single dose of C16TR for inhalation (Dose B) or matching placebo on Day 1 in Cohort 2.
  Interventions: Drug: C16TR; Drug: Placebo
- Cohort 3: C16TR Dose C or Placebo (Experimental): Participants were randomized to receive a single dose of C16TR for inhalation (Dose C) or matching placebo on Day 1 in Cohort 3.
  Interventions: Drug: C16TR; Drug: Placebo

INTERVENTIONS:
Drug: C16TR — Administered as inhalation using a Philips Micro device inhaler.
  Other Names: Hexadecyl-treprostinil
Drug: Placebo — Phosphate buffered saline (PBS) administered using Philips Micro device inhaler.
Drug: Tyvaso® — Administered as inhalation.
  Other Names: Inhaled treprostinil
  Arms: Cohort 1: Tyvaso®+C16TR Dose A or Tyvaso®+Placebo

SUMMARY:
The primary purpose of this study is to determine the safety and tolerability of escalating doses of C16TR for inhalation in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Have a body weight between 50 and 120 kg (females) or between 55 and 120 kg (males), inclusive, with a body mass index (BMI) between 19.0 and 32.0 kilograms per square meter (kg/m^2), inclusive, at screening.
* Have a medical history, physical examination, vital signs, electrocardiogram (ECG) and clinical laboratory results within normal limits or considered not clinically significant by the Investigator at screening.
* Do not take any systemic or topical prescription, or nonprescription (over-the-counter [OTC]) medication (acetaminophen or ibuprofen are permitted upon principal investigator [PI] discretion) within 2 weeks or 5 half-lives (whichever is longer) before first dose of the study drugs until discharge from the study (unless prescribed by the Investigator to treat an AE).
* Agree to abstain from consuming alcohol at least 3 days prior to in-clinic confinement until discharge from the study.

Exclusion Criteria:

* Have a history of anaphylaxis, a previous documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to any drug.
* Have a clinically significant history of neurological, cardiovascular, respiratory, endocrine, hematological, hepatic, renal, gastrointestinal, genitourinary, pulmonary, and/or musculoskeletal disease; glaucoma; a psychiatric disorder, or any other chronic disease, whether controlled by medication or not.
* Have a history of orthostatic hypotension, or unexplained syncope.
* Have a history of additional risk factors for Torsades de Pointes (eg, heart failure, family history of Long QT Syndrome).
* Are positive for human immunodeficiency virus (HIV) infection, hepatitis B surface antigen (HBsAg), or the hepatitis C virus (HCV) antibody at screening.
* Are users or former users of nicotine-containing products with > 10 pack-years of tobacco use history (including but not limited to cigarettes, cigars, and chewing or dipping tobacco), or users who stopped use or consumption (i.e., smoking, chewing, or pinching) of these nicotine-containing products less than 6 months before study drug administration or were using or had used topical or oral nicotine preparations for smoking cessation within the past 3 months before study drug administration.
* Have a history of alcohol abuse or a history of or current impairment of organ function reasonably related to alcohol abuse.
* Have a history or current evidence of abuse of licit or illicit drugs or a positive urine test for drugs of abuse.
* Have a history of abnormal bleeding tendencies.
* Donated any plasma within 7 days prior to first dosing, or has donated blood in excess of 450 mL, or had significant blood loss within 56 days prior to first dosing.
* Have any flu-like syndrome or other respiratory infection within 2 weeks of Day 1 or having been vaccinated with an attenuated live virus within 4 weeks of Day 1.
* Have a history of major surgery within 4 weeks or minor surgery within 2 weeks of screening.

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experienced an Adverse Event (AE) | Up to 32 days
  Safety and tolerability of escalating doses of C16TR for inhalation in healthy participants.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve (AUC) of Treprostinil and C16TR Post C16TR for Inhalation Dose | At multiple timepoints post dose on Days 2 to 4
Cohort 1: AUC of Treprostinil Post Tyvaso® Dosing | At multiple timepoints post dose on Days 1 and 2 for Cohort 1
  Pharmacokinetics of treprostinil after Tyvaso® dosing in healthy participants will be assessed.
Mean Change From Baseline in Corrected QT Interval by Fridericia (QTcF) for C16TR | Baseline up to Day 4 (Cohort 1) and Day 3 (Cohorts 2, 3, 4, and 5)

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://erj.ersjournals.com/content/48/suppl_60/PA2398.abstract